CLINICAL TRIAL: NCT03174665
Title: Incidence of Chronic Neuropathic Pain and Sensory Deficits After Nerve Repair Hand Surgery (Correlation With Genotypes and Biomarkers)
Brief Title: Chronic Neuropathic Pain After Nerve Repair Hand Surgery
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Uppsala University (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Adriana Miclescu, Associate professor, Uppsala University
Other Study IDs: ICONSS
Record Dates: First submitted 2017-05-30; First posted 2017-06-02 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Peripheral Nerve Injuries
MeSH Terms: conditions — Peripheral Nerve Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with Pain: Patients who had upper limb surgery or other trauma with a history of persistent spontaneous and/or evoked pain with duration of at least 3 months.
  Patients will be recruited to the study by using a postal follow up questionnaire. Patients who judge their pain at least moderate and/or affecting daily life by will be eligible and asked to participate. Patients will visit the Pain Clinic once. Oral and written information about the study will be provided, informed consent obtained. The affected nerve will be identified and the anatomy verified by ultrasound when needed.
  Interventions: Other: No intervention
- Patients with no pain: Patients operated with nerve suture surgery after a lesion of the nerves of upper extremity will be recruited to the study by using a postal follow up questionnaire. Patients with no pain will be asked to participate. Patients will visit the Pain Clinic once. Oral and written information about the study will be provided, informed consent obtained. The affected nerve will be identified and the anatomy verified by ultrasound when needed.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
This study intends to compare the patients with pain with those who underwent same procedure without developing pain. The patients with pain and without pain will be further analyzed in respect to clinical differences, biomarkers and genetical differences.

DETAILED DESCRIPTION:
Chronic pain is a well-known complication after surgery, but the prevalence of persistent pain after upper extremity surgery or other trauma affecting the radial, ulnar or the medial nerve, or branches of these nerves such as digital nerves is unknown. The reason that some patients develop persistent neuropathic pain after surgery, while others, who have been through the exact same procedure or trauma, are pain free is still unknown. The underlying mechanisms are still largely unknown. This can lead to different responses to treatment. Whenever possible, it is important to identify and address the underlying pain mechanisms in the individual patient in order to design an optimal treatment.

The aim of this study was to determine the prevalence and the factors implicated in the development of persistent pain after nerve suture surgery investigating Clinical symptoms, standardized clinical examination for neuropathic pain, 92 biomarkers special developed for neuropathic pain, genetics.

Conditioned pain modulation and Cold pressor test is intend to be performed in all the patients.

-

ELIGIBILITY:
Exclusion Criteria:

* Other condition that may confound assessment of pain attributed to posttraumatic upper limb pain, as judged by the investigator
* Any condition/disease that could interfere with the study measurements, e.g. peripheral vascular disease, diabetes mellitus, polyneuropathy etc as judged by the investigator

Inclusion Criteria:

* • Female or male subjects > 18 years of age

  * Provision of written informed consent
  * Be able to understand and comply with the requirements of the study
  * Patients with a history of persistent spontaneous and/or evoked pain (by e.g. touch, movement) interfering with daily activities of at least 3 months duration, associated with upper extremity surgery or other trauma affecting the radial, ulnar, medial or digital nerve
  * Spontaneous or evoked pain upon standardized test (mechanical, movement)> 50 on a 100 mm VAS scale in the group with pain after nerve repair surgery and a group of patients with no pain

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients opererated with nerve suture surgery on Hand Surgery between 2006-2014
Sampling Method: Non-Probability Sample
Enrollment: 990 (Actual)
Dates: Start 2016-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of neuropathic pain after trauma and nerve suture surgery | 2016 january-2017 january
  Patients with trauma and nerve suture surgery operated between 2006 and 2014 on Hand Surgery will receive a postal questionnaire (Leeds Assessment of Neuropathic Pain ). The patients with pain and without pain will be recruited to the study by using this postal follow up questionnaire. Patients who judge their pain at least moderate and/or affecting daily life by will be eligible and asked to participate.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Miclescu, MD, PhD, DEAA, Principal Investigator — Uppsala University Hospital

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Miclescu A, Ronngren C, Bengtsson M, Gordh T, Hedin A. Increased risk of persistent neuropathic pain after traumatic nerve injury and surgery for carriers of a human leukocyte antigen haplotype. Pain. 2024 Jun 1;165(6):1404-1412. doi: 10.1097/j.pain.0000000000003143. Epub 2023 Dec 22. PMID 38147413